CLINICAL TRIAL: NCT03357159
Title: A Phase II Study of Neovii Anti-human T-lymphocyte Immunoglobulin (ATLG, Grafalon®) With Post Transplant Escalated Doses of Post-transplant-Cyclophosphamide to Prevent Acute and Chronic GVHD Post Allogeneic Stem Cell Transplantation
Brief Title: Anti T-lymphocyte Immunoglobulin With Post Transplant Cyclophosphamide to Prevent GVHD Post Allogeneic Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof Arnon Nagler, M.D., M.Sc, Professor of Medicine Tel Aviv University, Director Hematology Division, Chair Israeli BMT Association,Chair of the ALWP of the EBMT, Co-Chair Scientific Council of the EBMT Chaim Sheba Medical Center, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-17-4055-AN-CTIL
Record Dates: First submitted 2017-10-09; First posted 2017-11-29 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Graft Versus Host Disease
Keywords: anti thymocyte globulin; cyclophospamide; graft-versus-host disease; stem cell transplantation
MeSH Terms: conditions — Graft vs Host Disease | interventions — Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: The patients will get conventional GVHD prophylaxis consisting of ATLG 15mg/kg total (5mg/kg day) on days -3 to -1 pre transplantation. Cyclophosphamide at 25mg/kg dose will be administrated at day +3 post infusion of the stem cell (SC) graft to the first 3 patients. If no > grade II toxicity* occurs, the next 3 patients will receive cyclophosphamide at 25mg/kg dose at day +3 and +4 post SC graft infusion. If no > grade II toxicity*occurs, the next 3 patients will receive cyclophosphamide at 37.5 mg/kg dose at day +3 and +4 post SC graft infusion. If no > grade II toxicity* occurs, the next 3 patients will receive the target dose of cyclophosphamide at 50 mg/kg dose on day +3 and +4 post SC graft infusion. The residual 18 patients will receive cyclophosphamide at the maximal tolerated dose (MTD) established in the first part of the study. Patients will also receive GVHD prophylaxis consisting of a cyclosporine and cellcept starting on day +5 after transplantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- cyclophosphamide and ATLG (Experimental): The study will include 2 phases. In the first phase escalated doses of post-transplant cyclophosphamide up to a maximal dose of 50 mg/kg administered on day +3 and +4 (target dose) will be added to a standard GVHD prophylaxis consisting of anti-human T-lymphocyte immunoglobulin (ATLG, Grafalon®, formerly ATG-Fresenius S, Neovii Pharmaceuticals) 15mg/kg total (5mg/kg day) on days -3 to -1 pre transplantation in order to find the maximally tolerated dose (MTD) of post-transplant cyclophosphamide (PTCy) in combination with pre-transplant immunosuppression by ATLG. The second phase will use the MTD cyclophosphamide dose identified in the first phase.
  Interventions: Drug: Cyclophosphamide; Drug: anti-human T-lymphocyte immunoglobulin (ATLG)

INTERVENTIONS:
Drug: Cyclophosphamide — In the first phase escalated doses of post-transplant cyclophosphamide up to a maximal dose of 50 mg/kg , the second phase will use the MTD cyclophosphamide dose identified in the first phase.
Drug: anti-human T-lymphocyte immunoglobulin (ATLG) — 15mg/kg total (5mg/kg day) on days -3 to -1 pre transplantation

SUMMARY:
Investigators hypothesize that combination of ATLG with PTCy in matched or mismatched unrelated hematopoietic stem cell transplantation will reduce acute and chronic GVHD incidence. Furthermore it will allow shortening of the length of post-transplantation immunosuppression with calcineurin inhibitor (CNI) administration (currently administrated in addition to ATG as GVHD prophylaxis in daily common practice)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MDS/AML
2. 18 years or older and willing and able to comply with the protocol requirements.
3. LVEF ≥ 40%. 2-D transthoracic echocardiogram (ECHO) is the preferred method of evaluation. Multigated Acquisition Scan (MUGA) is acceptable if ECHO is not available.
4. Patients undergoing 8-10/10 HLA matched unrelated and unmanipulated PBSC transplantation
5. Patients conditioned with reduced intensity or reduced toxicity conditioning of fludarabine with reduced dose (2 days) or myeloabalative doses (4 days) of busulfan or with treosulfan.
6. Patients must sign written informed consent.
7. Adequate birth control in fertile patients.

Exclusion Criteria:

1. Patients undergoing other type of transplantation or with other type of basic disease other than AML or MDS.
2. Patients with respiratory failure (DLCO < 30%).
3. Active congestive heart failure (New York Heart Association [NYHA] Class III to IV), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention.
4. Psychiatric conditions/disease that impair the ability to give informed consent or to adequately co-operate
5. Bilirubin > 3.0 mg/dl, transaminases > 3 times upper normal limit
6. Creatinine > 2.0 mg/dl
7. ECOG-Performance status > 2
8. Uncontrolled infection
9. Pregnancy or lactation
10. CNS disease involvement
11. Pleural effusion or ascites > 1 liter.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-06 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Overal survival | 24 months
  Overall survival will be calculated from the day of SCT until death or last follow-up. OS will be determined using Kaplan-Meyer product limit method.
Disease-free survival | 24 months
  Disease-free survival will be calculated from the day of SCT until relapse, death of any cause, or last follow-up. DFS will be determined using Kaplan-Meyer product limit method.

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Nagler, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No